CLINICAL TRIAL: NCT06906627
Title: Implementation pRogram to Improve Screening and Management for CKD in Diabetes (IRIS-CKD)
Brief Title: Implementation pRogram to Improve Screening and Management for CKD in Diabetes (Program 1) (IRIS-CKD)
Acronym: IRIS-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bayer (Industry); Boehringer Ingelheim (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00116493
Record Dates: First submitted 2025-02-21; First posted 2025-04-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease(CKD); Type 2 DM; Type 2 Diabetes Mellitus (T2DM)
Keywords: CKD; T2DM; T2D; Type 2 Diabetes; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: (IRIS-CKD Screening Program) is a randomized trial of delivery of a home testing kit for eGFR and/or UACR versus a standard laboratory order to increase rates of CKD screening in people who have lapsed beyond the recommended screening interval.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (IRIS-CKD Screening Program): Home Kit (Active Comparator): Home Kit: a kit delivered to participants home with instructions to complete eGFR (fingerstick) and/or UACR (urine sample) testing, depending on which lab(s) are missing at baseline.
  Interventions: Other: (IRIS-CKD Screening Program): Home Kit
- (IRIS-CKD Screening Program): Standard Lab Testing (Active Comparator): Standard Laboratory Testing: a traditional order will be placed into the Electronic Health Record (EHR) for eGFR and/or UACR testing, depending on which lab(s) are missing at baseline.
  Interventions: Other: (IRIS-CKD Screening Program): Standard Lab Order

INTERVENTIONS:
Other: (IRIS-CKD Screening Program): Home Kit — All participants approached for enrollment in Program 1 will receive National Kidney Foundational educational materials related to CKD screening in type 2 diabetes and study information. All enrolled participants will receive a message regarding study lab(s) results.
  Home Test Kit: a kit delivered to participants homes with instructions to complete eGFR (fingerstick) and/or UACR (urine sample) testing, depending on which lab(s) are missing at baseline.
  Arms: (IRIS-CKD Screening Program): Home Kit
Other: (IRIS-CKD Screening Program): Standard Lab Order — ll participants approached for enrollment in Program 1 will receive National Kidney Foundation educational materials related to CKD screening in type 2 diabetes and study information. All enrolled participants will receive a message regarding study lab
  Arms: (IRIS-CKD Screening Program): Standard Lab Testing

SUMMARY:
IRIS-CKD is an implementation study to improve guideline-recommended screening of chronic kidney disease (CKD) in individuals with type 2 diabetes (T2D) in the United States.

DETAILED DESCRIPTION:
IRIS-CKD Screening Program: will focus on CKD screening in T2D. We will identify patients with T2D that have not received appropriate screening for CKD within the last 15 months and randomize patients to receive either a home kit to complete CKD screening ("home kit") versus a standard laboratory order ("laboratory order"). The primary objective is to evaluate whether delivery of home testing kits versus standard laboratory testing influences the degree to which patients receive guideline-recommended CKD screening. Patients will complete approximately 3 months of follow-up.

ELIGIBILITY:
Screening Program-

Inclusion Criteria:

* Adults with type 2 diabetes (T2D)
* Receiving primary care within the healthcare system, Primary Care Provider (PCP) visit within the past 24 months (any PCP provider, including APP).
* Lack of estimated glomerular filtration rate (eGFR) and/or urine albumin- creatinine ratio (UACR) measurement in the prior 15 months within the EHR

Exclusion Criteria:

• Chronic kidney disease (CKD) diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
CKD Screening Lab Opportunity Score | 3 months
  Opportunity score of completion of missing guideline-recommended screening for CKD (eGFR and/or UACR) at 3 months.
  The opportunity score will be calculated as the ratio of the number of missing labs measured by month 3 divided by the number of missing labs at baseline.

SECONDARY OUTCOMES:
CKD Screening Lab Opportunity Score by Subgroup | 3 months
  Opportunity score across subgroups by missing baseline screening labs: UACR only, eGFR only, or both.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Pagidipati, MD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - University of Alabama, Birmingham, Alabama
  - University of Michigan, Ann Arbor, Michigan
  - Essentia Health, Duluth, Minnesota
  - Duke University, Durham, North Carolina
  - Baylor Scott & White, Temple, Texas

IPD SHARING:
Plan to Share IPD: No